CLINICAL TRIAL: NCT05443347
Title: Activity, Adiposity, and Appetite in Adolescents 2 Intervention
Acronym: AAAA2INT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robin Shook, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00002194; K01DK119545 (NIH)
Record Dates: First submitted 2022-06-17; First posted 2022-07-05 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Energy Balance; Appetite; Metabolism; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured exercise (Experimental): Adolescents randomized to the exercise will participate in a supervised structured exercise program (walking on a treadmill, cycling on a stationary bicycle, etc.) and expend an equivalent of 400 kcals/session (approximately 45-60 min/session) on three days/week. We will follow the protocol of Mentor Dr. Joseph Donnelly, with exercise prescriptions progressing from 150 kcal/session at intervention onset to reach the target exercise energy expenditure (EEEx) (400 kcal/session) at the end of month 3. EEEx will be assessed at baseline and monthly during the intervention to determine the duration of treadmill exercise required to achieve the EEEx goals. All supervised exercise will occur at the CCHLN on a treadmill with heart rate, speed, and grade monitored by an exercise specialist every five minutes.
  Interventions: Behavioral: Aerobic exercise
- Newsletter control (Active Comparator): Adolescents randomized to the newsletter control will receive with biweekly newsletters with "parenting tips, sample praise statements, and age-appropriate activities and recipes" identical to what has been used by others (Epstein et al., 2008), including existing group-based interventions with overweight/obese adolescents.
  Interventions: Behavioral: Newsletter

INTERVENTIONS:
Behavioral: Aerobic exercise — Supervised aerobic exercise
  Arms: Structured exercise
Behavioral: Newsletter — Biweekly newsletter
  Arms: Newsletter control

SUMMARY:
The objective of the study is to quantify the relationship between physical activity, metabolic function, and appetite in adolescents. To do this we will test our working hypothesis that high levels of regular moderate-to-vigorous physical activity (MVPA), as opposed to body weight status, results in a metabolic phenotype consisting of enhanced metabolic function and proper regulation of appetite. We will randomly assigning sedentary overweight/obese adolescents (N=44) to either a control or structured-exercise group for three months.

DETAILED DESCRIPTION:
he objective of the study is to quantify the relationship between physical activity, metabolic function, and appetite in adolescents. To do this we will test our working hypothesis that high levels of regular moderate-to-vigorous physical activity (MVPA), as opposed to body weight status, results in a metabolic phenotype consisting of enhanced metabolic function and proper regulation of appetite. We will randomly assigning sedentary overweight/obese adolescents (N=44) to either a control or structured-exercise group for three months.

Our study statistician Dr. Vincent Staggs will randomize participants after final eligibility is determined to either the newsletter control or exercise intervention, balanced by gender to ensure equal composition of males and females.

The sample size for Study 2 (Aim 2) was calculated based on data from our lab; a small pilot study with sedentary and active periods to test the feasibility of our laboratory protocols. Based on this preliminary data, which is similar to data in the existing literature, we estimate changes in appetite ratings (hunger) 11% from baseline, equating to effect sizes of 0.67, resulting in sample size calculations of N=35. Assuming a drop-out rate of 10% (n=4) during the three month intervention, which is typically observed in similar interventions conducted by Mentor Dr. Donnelly, final sample size is set at N=40.

Data analysis will be completed by the PI with assistance from the statistician Dr. Staggs and the mentorship team. For visual analog scale (VAS) appetite measures, which are assessed at multiple time points within a single measurement session, we will conduct analyses in two ways. First, we will conduct between group analyses using each of the seven individual assessments (e.g. 60 min post-meal) to see if the values differ by physical activity or body weight group. Second, we will also calculate area under the curve (AUC) for each variable of interest (e.g. hunger, ghrelin), and use that measure for the test of group differences. To address Aim 1, hypothesis 2, we will repeat the analyses described above and include insulin sensitivity as a covariate. To address Aim 2, hypothesis 3, we will conduct between group analyses of change over time using repeated measures ANOVA, using the same analysis techniques for the appetite variables as described in Aim 1 (single assessment and AUC), with insulin sensitivity included as a covariate.

Appetite is considered the primary outcome of Aim 1 and 2. Subjective assessment of hunger and palatability will be completed using self-rated visual analogue scales (VAS), with each scale consisting of a 10-cm long line separating statements such as ?not at all hungry? and ?extremely hungry?. Perceptions of dietary restraint, disinhibition, and hunger will be measured during each measurement session prior to the fixed meal using the Three Factor Eating Questionnaire (TFEQ). The Control of Eating Questionnaire (CEQ) will be used to assess hunger, fullness, cravings, the desire to eat certain types of foods, and the ability to resist urges to eat. Objective assessment of appetite will be completed using blood samples taken from an indwelling catheter, and analyzed for episodic regulation of the following fasting and satiety hormones: glucose, insulin, leptin, ghrelin, glucagon-like peptide 1 (GLP-1), and peptide YY (PYY). All samples will be mixed a standard preservative (400 ?L of 10,000 KIU aprotinin), centrifuged, the plasma divided into aliquots and stored in -80?C freezer until analysis using standard kits at an outside certified clinical laboratory.

Appetite measured will be assessed following a fixed standard breakfast (40% of RMR, composed of 55% carbohydrate, 15% protein, 30% fat). The fixed breakfast will be administered while the participant is in a fasted state (?12 hours since last meal) and they will be asked to consume the meal within 15 minutes. Food intake (total kcals) will be assessed using an ad libitum pizza meal served three hours after the fixed meal. Participants will be instructed to eat until comfortably full and informed that they can request more of the meal at any point. Meals will be provided in 400 kcal portions, and each bowl of food will be weighed before and after serving, without the subjects? knowledge, and the amount consumed recorded. All meals will be served in a quiet dining room free from distractions located at CCHLN. All foods will be prepared using a standard procedure in the metabolic kitchen to ensure consistency across the treatment conditions, and nutrient composition of the meals will be determined using nutrient analysis software (Nutrient Data System for Research, version 2016).

Insulin sensitivity via the euglycemic ?hyperinsulinemic clamp technique is considered the primary outcome for Aim 1, hypothesis 2. Participants will arrive fasted (12-hours overnight). A catheter will be inserted into an antecubital vein of one arm to infuse insulin and 20% dextrose, and another catheter will be inserted into the contralateral antecubital vein for blood sampling. The participant will rest quietly and RQ via indirect calorimetry will be measured (see Resting Metabolic Rate), followed by collection of 3 baseline blood samples to establish baseline glucose levels. Immediately following and lasting for 180 minutes, a primed continuous infusion of regular human insulin will be administered at a rate of 40 mU?m2 body surface area?1?min?1 along with a variable infusion of 20% dextrose to maintain euglycemia to match baseline levels (expected 90-100 mg/dL). Blood glucose measurements will be completed every five minutes for determination of glucose infusion rate using a YSI-2300 analyzer. Furthermore, every ten minutes blood will be drawn into serum separator tubes, centrifuged, and stored at -80? C for later insulin analysis. RQ will again be measured 2 hours into the clamp for a period of 15 minutes. Insulin sensitivity will be determined by the glucose disposal rate during the final 45 min of the hyperinsulinemic-euglycemic clamp when euglycemia has been established. This procedure will occur at the KUMC Clinical and Translation Science Unit research facility.

Adolescents will be randomly assigned to either an exercise or newsletter control condition for three months. Adolescents randomized to the exercise will participate in a supervised structured exercise program (walking on a treadmill, cycling on a stationary bicycle, etc.) and expend an equivalent of 400 kcals/session (approximately 45-60 min/session) on three days/week. We will follow the protocol of Mentor Dr. Joseph Donnelly, with exercise prescriptions progressing from 150 kcal/session at intervention onset to reach the target exercise energy expenditure (EEEx) (400 kcal/session) at the end of month 3. The rationale for this dose of structured exercise is based on national and international physical activity recommendations for youth of 60 minutes/day, along with data from the Donnelly team and others that indicates this level of exercise over a three month period will result in improvements in cardiorespiratory fitness in adolescent participants.

EEEx will be assessed at baseline and monthly during the intervention to determine the duration of treadmill exercise required to achieve the EEEx goals. EEEx will be assessed by indirect calorimetry (TrueOne 2400 Metabolic Measurement Cart, ParvoMedics, Salt Lake City, Utah) at one minute intervals. The Weir equation will be used to calculate EEEx from measured oxygen consumption and carbon dioxide production. Prior to each EEEx assessment participants will perform a brief warm-up (~ 2 minute, 3?4 mph, 0% grade). At the baseline assessment, treadmill speed/grade will begin at 3 mph/0% grade and will be adjusted by increments of 0.5 mph/1% grade until the participant reaches 70% HR max ?4 beats/minute. At the end of months 1 to 3, EEEx will be calculated at both 70% and 80% of heart rate (HR) maximum to accommodate personal preferences for walking or running. EEEx will be assessed at both 70% (15 minutes) and 80% HR max (15 minutes) with a 2 minute interval between assessments to allow participants to remove the mouthpiece and obtain water if desired. Either speed or grade will be adjusted depending on participant preference. The average EEEx over a 15 minute interval (kcal/minute) will be used determine the duration of exercise sessions performed during the first month. For example: EEEx = 9.2 kcal/minute, prescribed exercise = 400 kcal/session, exercise duration = 400/9.2 = 44 minutes/session.

All supervised exercise will occur at the CCHLN on a treadmill with heart rate, speed, and grade monitored by an exercise specialist every five minutes. Televisions and iPads will be available for the participants to watch while exercising. Compliance will be defined as completion of ?90% of scheduled exercise sessions/week and participants will be excluded if they fail to meet this requirement. Successful completion of an exercise session will be defined as maintaining target HR ?4 beats/minute for the prescribed exercise duration.

As has been done in previous studies by pediatric obesity treatment experts we will use a newsletter control group. Just as in these previous studies, families will receive a monthly newsletter with ?parenting tips, sample praise statements, and child-appropriate activities and recipes? identical to what has been used in the work of leaders in the field of pediatric obesity. The content will be similar to that delivered in existing group based interventions with overweight/obese adolescents at the CCHLN under the direction of Mentor Dr. Ann Davis.

Energy intake will be assessed using three methods: 1) objectively, as measured by amount of kcals consumed during an ad libitum meal (see above, section Fixed/Ad libitum meals), 2) subjectively, assessed in each free-living 7-day assessment period via dietician-administered 24-hour dietary recalls, and 3) calculated, based on intake-balance method. Subjective energy intake will be assessed using three dietary recalls occurring on randomly selected non-consecutive days over each 7-day free-living assessment period (including at least one weekend day) to minimize preparation that could bias recall, by a team of experienced (>6 years using Nutrient Data System for Research software) registered dietitians employing a multi-pass approach, which utilizes prompting to reduce food omissions and standardizes the interview methodology across interviewers. Estimated energy intake will also be calculated using the intake-balance method during each treatment condition, based on the principles of the First Law of Thermodynamics, using the following equation: calculated energy intake= 1,020 (?FFM/?t) + 9,500(?FM/?t) + EE, where ?FFM and ?FM represent change in each variable as measured by DXA at the beginning and end of each assessment period condition, ?t represents days between measurements; 1,020 and 9,500 represent the energy density in kcals of FFM and FM per kg, respectively; and EE represents energy expenditure as measured by the activity monitor.

Energy expenditure will be estimated during each 7-day free-living assessment period using an arm-based monitor (SenseWear Mini?, BodyMedia Inc.), which calculates energy expenditure using tri-axial accelerometry and measures of heat flux, galvanic skin response, skin temperature, and near-body ambient temperature.

Body composition including fat mass and fat-free mass will be measured using a whole-body dual energy X-ray absorptiometer (DXA, Lunar DPX system, version 3.6) with the participant dressed in surgical scrubs and in bare feet.

ELIGIBILITY:
Inclusion Criteria:

* Tanner Stage III-V, as determined via self-assessment
* Non-smoking
* Not currently involved in any other research study
* No meds that may alter metabolism
* Sedentary (<60 min/day exercise)
* Willing to participate in an exercise program

Exclusion Criteria:

* BMI <5th percentile or >99th percentile for age and sex
* Weight not stable
* Restrained eater (>13 on the restraint section of the three-factor eating questionnaire; Current/past diagnosis of an eating disorder.
* Self-reported medical conditions (including, but not limited to, diabetes, Crohn's disease, etc.) that may affect adherence to the protocol, exercising safely, or alter metabolism
* Taking medications know to affect metabolism (e.g. thyroid medication, β-blockers, or stimulants).
* Gave birth in the past 12 months or <6 months post-lactation.
* Active (>60 min/day exercise)
* Not willing to participate in an exercise program

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin P Shook, PhD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated results will be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Structured Exercise | Newsletter Control
Started | 19 | 12
Completed | 14 | 11
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Structured Exercise | Newsletter Control | Total
Number analyzed (Participants) | 19 | 12 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 12 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (1.1) | 15.6 (0.9) | 15.9 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 15 | 8 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Appetite- Subjective
Description: The investigators will measure subjective appetite ratings using visual analog scales related to hunger following a fixed-calorie meal: Hunger, Area Under the Curve (AUC)
  Hunger and palatability were assessed using self-rated visual analogue scales (Rogers, P. J., & Blundell, J. E. (1993). Intense sweeteners and appetite. The American Journal of Clinical Nutrition, 58(1), 120-122.) Scale is 0-100, with 0 equaling 'I am not hungry at all' and 100 equaling 'I have never been more hungry'.
  Area under the curve (AUC) was calculated for appetite variables by calculating the area of the response as you would a trapezoid.
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: score*minute
Arm/Group | Structured Exercise | Newsletter Control
Number analyzed (Participants) | 14 | 11
score*minute | 6282 (1075) | 8738 (1171)

2. Primary Outcome: Appetite- Objective
Description: he investigators will measure objective appetite responses using plasma ghrelin following a fixed-calorie meal.
Time Frame: 3 months
Population: Plasma ghrelin values were not assessed. Blood samples needed for assessment were not obtained due to lack of staff. Samples will not be collected in the future.
Arm/Group | Structured Exercise | Newsletter Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Appetite- Adjusted
Description: The investigators will measure objective and subjective appetite responses as described above adjusted by insulin sensitivity (glucose infusion rate, mg/kg/min) as assessed in the euglycemic hyperinsulinemic clamp technique.
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale*min
Arm/Group | Structured Exercise | Newsletter Control
Number analyzed (Participants) | 14 | 11
score on a scale*min | 7482 (1094) | 8269 (1094)

ADVERSE EVENTS:
Time Frame: Average of 117 days
Arm/Group | Structured Exercise | Newsletter Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/12
Other Adverse Events (participants affected / at risk) | 0/19 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Structured Exercise (N=19) | Newsletter Control (N=12)
Sore arm following IV (General disorders) | 0 (0) | 1 (1) — Sore arm following IV placement
Skin reaction to activity monitor (General disorders) | 0 (0) | 1 (1) — Skin reaction to wearing activity monitor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT05443347/Prot_SAP_000.pdf